CLINICAL TRIAL: NCT03475888
Title: Incidence of Ventricular Arrhythmias in Patients With Chronic Total Occlusion Recanalization
Acronym: VACTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Sing-Chien Yap, MD, PhD, Principal investigator, Erasmus Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL59827.078.16
Record Dates: First submitted 2018-03-12; First posted 2018-03-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: Chronic Total Occlusion of Coronary Artery; Ventricular Arrythmia; Sustained VT; Ventricular Fibrillation; Implantable loop recorder
MeSH Terms: conditions — Ventricular Fibrillation

STUDY DESIGN:
Intervention Model Description: Single center pilot study of patients with CTO.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Patients who have undergone a successful percutaneous CTO recanalization
  Interventions: Device: Medtronic Reveal LINQ™ Insertable Cardiac Monitor (ICM)
- Group B (Active Comparator): Patients who have undergone a failed percutaneous CTO recanalization or have an untreated CTO
  Interventions: Device: Medtronic Reveal LINQ™ Insertable Cardiac Monitor (ICM)

INTERVENTIONS:
Device: Medtronic Reveal LINQ™ Insertable Cardiac Monitor (ICM) — Implantation of Medtronic Reveal LINQ™ ICM

SUMMARY:
A chronic total occlusion (CTO) is common in patients with coronary artery disease. CTO recanalization has been shown to improve survival in comparison to failed CTO recanalization. Whether this is related to ventricular arrhythmias (VA) is unknown. The purpose of this pilot study is to evaluate the incidence of VA after successful CTO recanalization and in those with failed CTO recanalization or untreated CTO. Patients will be monitored using an insertable cardiac monitor.

DETAILED DESCRIPTION:
Rationale: Successful chronic total occlusion (CTO) recanalization has been associated with improved long-term survival. Furthermore, CTO is an independent predictor for the occurrence of ventricular arrhythmias (VA) in patients with ischemic cardiomyopathy and implantable cardioverter defibrillators (ICDs). One may speculate that a successful CTO recanalization may provide electrical stability. However, no data are available on the incidence of sustained VA in this patient population.

Objective: The objective of the present pilot study is to assess the incidence of sustained VA in 2 CTO groups: patients with successful percutaneous CTO recanalization (group A), patients with failed percutaneous CTO recanalization or untreated CTO (group B).

Study design: Pilot study of patients with CTO.

Study population: A total of 90 patients will be enrolled with a maximum of 45 patients in each arm.

Intervention: A Medtronic Reveal LINQ™ Insertable cardiac monitor (ICM) will be implanted in every patient to continuously monitor heart rhythm during the follow-up period.

Main study parameters/endpoints: To assess the incidence of VA defined as sustained ventricular tachycardia >30 s or ventricular fibrillation.

ELIGIBILITY:
Inclusion criteria:

1. Presence of CTO defined as complete obstruction of the vessel with Thrombolysis In Myocardial Infarction (TIMI) flow grade 0 and an estimated duration of ≥3 months, and one of the following:

   1. A successful percutaneous CTO recanalization for stable angina within the previous 6 months. A successful CTO recanalization is defined as a final TIMI flow grade ≥2 and a residual stenosis ≤30% after stent implantation.
   2. A failed percutaneous CTO recanalization for stable angina within the previous 6 months. A failed CTO recanalization is defined as not fulfilling the criteria for successful CTO recanalization.
   3. Untreated CTO diagnosed in the previous 6 months.
2. Age ≥18 years.
3. Written informed consent.
4. Patient agrees to the follow-up including the implantation of the ICM.

Exclusion Criteria:

1. Patients who are potential candidates for an ICD according to the 2015 ESC guidelines.
2. Patients who have a cardiac implantable electrical device (CIED) (e.g., pacemaker, ICD).
3. Patient has reduced immune function or is otherwise at high risk for infection.
4. Patient has had a recent (within 30 days) or otherwise unresolved infection.
5. Known pregnancy at time of inclusion.
6. Patient has severe co-morbidity that may cause the patient to be non-compliant with the protocol, confound the data interpretation or is associated with limited life expectancy (i.e., less than one year).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Ventricular Arrhythmias | 3 years after ICM implantation
  Sustained ventricular tachycardia (>30 s) or ventricular fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Sing-Chien Yap, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - VUMC, Amsterdam
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Assaf A, Sakhi R, Diletti R, Hirsch A, Allaart CP, Bhagwandien R, Firouzi M, Smits PC, Hoogendijk MG, Theuns DAMJ, Yap SC. Incidence of ventricular arrhythmias in patients with chronic total coronary occlusion: Results of the VACTOR study. Int J Cardiol Heart Vasc. 2023 Dec 18;50:101323. doi: 10.1016/j.ijcha.2023.101323. eCollection 2024 Feb. PMID 38188347